CLINICAL TRIAL: NCT05708508
Title: Effectiveness of an Immune-guided Cytomegalovirus Infection Preventive Strategy Compared to a Universal Prophylactic Strategy in Renal Transplant Patients
Acronym: CYTOPREV
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020/0422/HP
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Kidney Transplant Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Immuno-guided strategy" arm (Experimental): * Patients in the "low risk" group will be monitored between D+15 and W+28 according to a strategy preemptive.
  * Patients in the "high risk" group (anti-CMV response <130 SFC/106 cells) will be treated according to the terms of the "universal prophylaxis" arm from D+15 and until W+15.
  At the W+15 visit:
  * If the patient is considered at "low risk", the antiviral treatment is stopped and he will continue the follow-up according to the modalities of the "universal prophylaxis" arm until W+28.
  * If the patient is still at "high risk" antiviral treatment will be continued until W+28.
  Interventions: Drug: ROVALCYTE
- "Universal prophylaxis" arm (Active Comparator): Patients will receive from D+15 post-transplant an antiviral treatment with valganciclovir (ROVALCYTE) for the first 3 months following the transplant. Clinico-biological monitoring during the 6 months according to the usual practices of the 2 centers and monitoring of CMV DNAemia.
  Interventions: Drug: ROVALCYTE

INTERVENTIONS:
Drug: ROVALCYTE — "Immuno-guided strategy" arm

SUMMARY:
Cytomegalovirus (CMV) establishes a chronic infection in 60% of the general population. In renal transplant recipients, it is responsible for morbidities occurring mainly in the first 6 months after transplantation. These include viral reactivations linked to immunosuppressive treatment inhibiting the anti-CMV T lymphocyte response. CMV infection, a sign of uncontrolled viral replication, is defined by the detection of viral DNA in the peripheral blood (DNAemia). CMV disease is defined as the association of an infection and symptoms attributable to the virus.

In transplant recipients carrying the virus before transplantation (positive serology: CMV+), two infection prevention strategies are recommended: either close monitoring of DNAemia with antiviral treatment in the event of positive detection (pre-emptive strategy), or antiviral treatment for the first 3 months following the transplant (prophylactic strategy). Both strategies result in the occurrence of CMV infection in 15 to 20% of patients within the first 6 months, with the majority of events occurring between 3 and 6 months.

Numerous studies show that the evaluation of the anti-CMV T lymphocyte response, either before (D0) or early after transplantation (D15), or when antiviral prophylaxis is stopped, allows the identification of patients at risk of CMV infection. No study has yet demonstrated the contribution of such an evaluation in a preventive strategy. We therefore propose such a study.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patient for 1 to 12 days
* CMV seropositivity on the day of transplantation: IgG threshold =6 AU/mL CMIA CMV IgG, Architect i4000 (Abbott)) (Serology performed on D0, before the transplant)
* Non-depleting inducing immunosuppressive treatment (Basiliximab) (implementation before the transplant)
* Affiliation to a social security scheme
* Patient having read and understood the information letter and signed the consent form

Exclusion Criteria:

* Active CMV infection (detectable CMV DNAemia - peripheral CMV DNAemia ≥ 305 IU/mL)
* Patient with hypersensitivity to valganciclovir, ganciclovir, aciclovir or valaciclovir or to any of the excipients
* Lympho-depleting inducing immunosuppressive treatment (antithymoglobulins)
* Neutropenia (neutrophils < 500/mm3) or thrombocytopenia (platelets < 25,000/mm3) or anemia (hemoglobin < 8G/L) identified on routine care samples taken on the day of inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate, in CMV+ transplant patients, the efficacy of an immuno-guided preventive strategy compared to the universal prophylactic strategy, in terms of CMV infection in the 6 months following kidney transplantation. | 6 months
  Proportion of patients with CMV infection within 6 months of transplantation.

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668